CLINICAL TRIAL: NCT00314626
Title: Multicentre, Open Label, Prospective, Randomised Clinical Trial of an Antiretroviral Simplification Treatment With Efavirenz + Abacavir + 3TC Once Daily
Brief Title: Antiretroviral Treatment Simplification Study With Efavirenz + Abacavir + 3TC Once Daily
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: LLuita Sida Foundation, LLuita Sida Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELA; 2004-001198-25
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2007-11

CONDITIONS: HIV Infections
Keywords: Antiviral efficacy; Tolerability; Immunologic response; Virologic response; HIV
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): abacavir 600 mg + lamivudine (3TC) 300 mg in 1 tablet + efavirenz 600 mg 1/24h
  Interventions: Drug: efavirenz; Drug: Abacavir+lamivudine
- B (No Intervention): efavirenz + 2 NUCS

INTERVENTIONS:
Drug: efavirenz — Efavirenz
  Other Names: sustiva
  Arms: A
Drug: Abacavir+lamivudine — Abacavir+lamivudine
  Other Names: Kivexa
  Arms: A

SUMMARY:
To evaluate the proportion of patients with virological failure after 48 weeks of treatment with the combination of efavirenz 600 mg + lamivudine (3TC) 300 mg + abacavir 600 mg once daily as an antiretroviral simplification regimen.

DETAILED DESCRIPTION:
Treatment simplification is a therapeutic strategy that allows patients with controlled viral replication to switch to an easier-to-take antiretroviral system to promote long-term adherence and thus maintain controlled viral load for longer, delaying the evolution of the HIV infection.

The combination of ABC+3TC+EFV is a potent and easy-to-take regimen (2 tablets once a day) that could be suitable for the simplification of antiretroviral treatment in patients with controlled viral load with a regimen that includes 2 NRTI taken twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. HIV-1 infected patients.
3. Patients on HAART therapy including efavirenz and two NRTIs in a twice-daily regimen for 6 months at least.
4. Patients with an undetectable HIV-1 viral load over the last 6 months (at least 2 determinations separated by 3 months).
5. Subject able to follow the treatment period.
6. Signature of the informed consent.
7. Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use a barrier contraceptive method during the study.

Exclusion Criteria:

1. Hepatic tests > 5 times above normality.
2. Pregnancy or breastfeeding
3. Presence of opportunistic infections and/or recent tumours (< 6 months).
4. Suspected or documented resistance to any of the investigational drugs.
5. Known allergic hypersensitivity to any of the investigational drugs or any similar drug.
6. Subjects with abusive consumption of alcohol or illegal drugs.
7. Patients participating in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Viral load of HIV-1 at each visit with regard to the baseline visit. | At 12, 24, 36 and 48 weeks

SECONDARY OUTCOMES:
To evaluate immunological efficacy (changes in the CD4 and CD8 counts) of the combination studied over the follow-up period. | At 12, 24, 36 and 48 weeks
To evaluate the tolerance and safety of the combination of abacavir+ lamivudine (in a single tablet) + efavirenz given once daily over 48-week treatment period. | At 12, 24, 36 and 48 weeks
To evaluate treatment adherence (assessed by a self-reported questionnaire and with graduated satisfaction scales) and patient quality of life (assessed by means of the MOS-HIV questionnaire). | At 12, 24, 36 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD, PhD, Principal Investigator — Lluita contra la Sida Foundation-HIV Unit
Locations (16):
- Spain (16):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital de la Vall d'Hebron, Barcelona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital de Aranzazu, Donostia / San Sebastian, Guipuzcoa
  - Hospital San Millan de Logroño, Logroño, La Rioja
  - Hospital Arnau de Vilanova de Lleida, Lleida, Lleida
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Severo Ochoa Leganés, Madrid, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Cristal-Piñor, Ourense, Ourense
  - Hospital Santa María Nai, Ourense, Ourense
  - Hospital de Navarra, Pamplona, Pamplona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital General de Valencia, Valencia, Valencia